CLINICAL TRIAL: NCT01083472
Title: A Multicenter, Prospective, Single-Blind, Randomized, Controlled Study of the Repair of Challenging Abdominal Wall Defects: Strattice(TM) TM in Abdominal Wall Repair
Brief Title: Repair of Challenging Abdominal Wall Defects: Strattice(TM) TM in Abdominal Wall Repair (StAR)
Acronym: StAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Surgical practice evolution changed acceptable standard of care and lead to potential enrollment bias.
Sponsor: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LFC2009.01.01
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-09

CONDITIONS: Hernia; Surgical Wound Dehiscence
Keywords: dehiscence; laparotomy; Hernia repair; surgical wound; surgical mesh
MeSH Terms: conditions — Hernia; Surgical Wound Dehiscence; Surgical Wound | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strattice(TM) TM repair (Active Comparator): Strattice(TM) TM will be placed in the intraperitoneal or retrorectus position to support the repair of abdominal wall defect
  Interventions: Device: Strattice(TM) Reconstructive Tissue Matrix
- Standard of Care repair (Active Comparator): Abdominal wall defect will be repaired using current standard of care techniques of either suture alone or suture with absorbable surgical mesh
  Interventions: Procedure: Suture/suture with absorbable mesh

INTERVENTIONS:
Device: Strattice(TM) Reconstructive Tissue Matrix — Strattice(TM) TM will be used to support the repair of abdominal wall defect
  Arms: Strattice(TM) TM repair
Procedure: Suture/suture with absorbable mesh — Abdominal wall defect will be repaired with suture alone or absorbable mesh with suture
  Arms: Standard of Care repair

SUMMARY:
The objective of this study is to compare the incidence of post-repair wound related complications, including hernia occurrence/recurrence, between challenging abdominal wall defects repaired with Strattice(TM) Reconstructive Tissue Matrix (TM) and those managed by standard repair. It is hypothesized that the use of Strattice(TM) TM to reinforce the repair will reduce the incidence of these post-repair complications.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-blind, randomized, longitudinal, cross-over evaluation of the repair of challenging abdominal wall defects using Strattice(TM) TM or standard surgical repair. These abdominal wall defects can be acute or chronic, and include midline, transverse (including flank) as well as Pfannenstiel incisions. The skin may be closed (fascial dehiscence or incisional hernia) or open (patient with open abdomen or acute fascial dehiscence) with or without evisceration. Patients randomized to the control group who require a re-operation to perform the planned final repair or due to failure of the initial repair within 12 months, will be offered repair with Strattice™ TM (i.e. "crossed over") or if such repair not performed, the patient will have completed the study. An adaptive study design will be used to validate the initial conditional power of the study and a balanced randomization, based upon the three conditions (type of defect [dehiscence, hernia repair or open abdomen], morbidity [POSSUM score] and time since exposure of abdominal fascia/viscera) will be used to equally distribute subjects between groups.

The primary endpoint of this study is hernia occurrence at 12 months post repair and secondary endpoints include re-operation for abdominal wall repair within 12 months, incidence of complications requiring intervention(medical or surgical) within the first 30 days after repair,, length of hospitalization and resource utilization, and all cause mortality.

Subjects will be enrolled and randomized to receive Strattice(TM) TM reinforcement of repair or standard of care repair (i.e. suture alone or suture with absorbable mesh) and followed at set timepoints to observe incision site repair for surgical site events, including reoperation and hernia occurrence.

ELIGIBILITY:
Inclusion Criteria:

* adults (18years of age or older) who is able to provide written informed consent for study participation
* has need of surgical intervention for repair of (potentially) contaminated abdominal wall defect of >3cm and <22cm in length, where the viscera have not been exposed for more than 15 days in case of open abdomen(skin and fascia open).
* Is willing and able to return for all scheduled & required study visit.

Exclusion Criteria: at the time of randomization

* severe systemic sepsis
* frank pus in the wound, a fistula that will not be closed at the time of surgery or intra-abdominal abscess in surgical area,
* ongoing necrotizing pancreatitis,
* Is on chronic immunosuppressive therapy, or other medication that influences wound healing
* requires only short-term temporary closure,
* requires a synthetic, non-absorbable mesh to close the abdominal wall defect
* is unable to undergo general anesthesia,
* has other major organ system dysfunction or disorder that would jeopardize subject completing the 24 month study.
* Is unable to undergo an MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angus JM Watson, Principal Investigator — Raigmore Hospital, Inverness Scotland, National Health Service, UK; Berndt Reith, Principal Investigator — Klinikum Konstanz, Konstanz Germany; Johannes Jeekel, Study Chair
Locations (29):
- France (3):
  - CHU Amiens Hopital Nord, Amiens
  - Hopital de la Pitie-Salpetriere, Paris
  - CHU Robert Debre, Reims
- Germany (16):
  - Universitätsklinikum Aachen, Aachen
  - Unfallkrankenhaus Berlin, Berlin
  - St. Josef-Hospital, Bochum
  - Kliniken der Stadt Köln, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum und Fachbereich Medizin der Johann Wolfgang Goethe Universitat, Frankfurt am Main
  - Universitätsklinikum Giessen und Marburg GmbH, Giessen
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Krankenhaus Agatharied GmbH, Hausham
  - Krankenhaus Salem der Evang. Stadtmission Heidelberg, Heidelberg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Klinikum Konstanz, Konstanz
  - LMU Klinikum der Universität München, München
  - Technischen Universität München - Klinikum rechts der Isar, München
  - Lukaskrankenhaus, Neuss
  - Klinikum St Elisabeth Straubing GmbH, Straubing
- St Orsola-Malpighi University Hospital, Bologna, Italy
- Netherlands (3):
  - Academisch Ziekenhuis Maastrict, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - Haga Ziekenhuis, The Hague
- Hospital Universitari del Mar, Barcelona, Spain
- United Kingdom (5):
  - Sandwell General Hospital, Birmingham
  - Raigmore Hospital, Inverness
  - Manchester Royal Infirmary, Manchester
  - Heart of England NHS Trust, Solihull
  - Arrowe Park Hospital, Upton, Wirral

REFERENCES:
- [Background] Van Geldere D. One hundred years of abdominal wound dehiscence and nothing has changed. Hernia 2000; 4:302-4.
- [Background] van't RM, De Vos Van Steenwijk PJ, Bonjer HJ, Steyerberg EW, Jeekel J. Incisional hernia after repair of wound dehiscence: incidence and risk factors. Am Surg. 2004 Apr;70(4):281-6. PMID 15098775
- [Background] Murugappan K, Gomes F, Waxman B. Abdominal wound dehiscence - who is really at risk? ANZ J Surg 2009; 79(S1):A25
- [Background] Gislason H, Viste A. Closure of burst abdomen after major gastrointestinal operations--comparison of different surgical techniques and later development of incisional hernia. Eur J Surg. 1999 Oct;165(10):958-61. doi: 10.1080/110241599750008071. PMID 10574104
- [Background] Webster C, Neumayer L, Smout R, Horn S, Daley J, Henderson W, Khuri S; National Veterans Affairs Surgical Quality Improvement Program. Prognostic models of abdominal wound dehiscence after laparotomy. J Surg Res. 2003 Feb;109(2):130-7. doi: 10.1016/s0022-4804(02)00097-5. PMID 12643854

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Strattice(TM) TM Repair | Standard of Care Repair
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Strattice(TM) TM Repair | Standard of Care Repair | Total
Number analyzed (Participants) | 18 | 19 | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 70 (9.94) | 67 (8.49) | 68.5 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Hernia Occurrence
Description: Hernia occurrence will be assessed by clinical evaluation. At Month 12 and at any time during the study if hernia occurrence is clinically suspected, a magnetic resonance image (MRI) will be obtained.
Time Frame: Month 12 after repair
Population: Due to early termination of the study and the low enrollment number (only 37 subjects out of the planned 200 subjects being enrolled), all planned analyses of study endpoints were not performed. The only study results obtained focused on safety. Due to the small sample size these safety results should be interpreted with caution.
Arm/Group | Strattice(TM) TM Repair | Standard of Care Repair
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Strattice(TM) TM Repair | Standard of Care Repair
Serious Adverse Events (participants affected / at risk) | 7/18 | 8/19
Other Adverse Events (participants affected / at risk) | 16/18 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strattice(TM) TM Repair (N=18) | Standard of Care Repair (N=19)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infectious Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Post Operative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 3 (3) | 1 (1)
Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Dehiscence (Infections and infestations) | 3 (3) | 7 (8)
Wound Necrosis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound Secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Circulatory Collapse (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strattice(TM) TM Repair (N=18) | Standard of Care Repair (N=19)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Cardiac Disorders (Cardiac disorders) | 1 (1) | 1 (1)
Endocrine Disorders (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal Disorders (Gastrointestinal disorders) | 5 (5) | 7 (7)
General Disorders Administration Site Conditions (General disorders) | 3 (3) | 4 (4)
Infections and Infestations (Infections and infestations) | 11 (11) | 9 (9)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 9 (9) | 12 (12)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nervous System Disorders (Nervous system disorders) | 2 (2) | 0 (0)
Renal and Urinary Disorders (Renal and urinary disorders) | 1 (1) | 1 (1)
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Surgical and Medical Procedures (Surgical and medical procedures) | 1 (1) | 0 (0)
Vascular Disorders (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other